CLINICAL TRIAL: NCT05601297
Title: Acceptability of Women to Intimate Partner Violence and Its Correlates Among Attendants of Maternal and Child Health Center in Assiut City
Brief Title: Acceptability of Women to Intimate Partner Violence and Its Correlates Among Attendants of Maternal and Child Center in Assiut
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hagar Ahmed Abdel Hameid, doctor, Assiut University
Other Study IDs: partner violance against women
Record Dates: First submitted 2022-10-24; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Violence Against Women

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questationair — acceptability of women to partner violance

SUMMARY:
identify acceptability of ever married women against intimate partner violence and its correlates among women attending primary health care in Assiut city.

DETAILED DESCRIPTION:
Violence against women is a major public health problem . World Health Organization estimates that globally 30% of women have been subjected to either physical and/or sexual intimate partner violence(IPV) or non-partner sexual violence in their lifetime.

IPV refers to any behaviour within an intimate relationship that causes physical, psychological or sexual harm to those in the relationship. IPV definition covers violence by both current and former spouses and partners. Forms of intimate partner violence include: Acts of physical violence, sexual violence, emotional (psychological) abuse, and controlling behaviors.

Initial studies on IPV against women tended to concentrate on assessment of incidence and prevalence. Although prevalence is critical, reducing or eliminating some problems also requires comprehension of cultural norms and expectations.

An ecological approach showed that public attitudes accepting or justifying violence and aggression are a risk factor at a macro social level, as they can encourage or deter its occurrence in societies.

UN Women reported that among Egyptian women in reproductive age, the prevalence of lifetime physical and/or sexual intimate partner violence was 26% and the prevalence of physical and/or sexual intimate partner violence in the last 12 months was 14 %.

The Egyptian studies that assessed attitudes of acceptability of IPV and their predictors has explored acceptability to only one form of IPV. Using a single-item measures, they measured justification for the husband's use of more severe physical force in response to the wife's violation of expected domestic roles or his patriarchal control in marriage.

ELIGIBILITY:
Inclusion Criteria:

* Ever married women (current married women and who were married since one year) who seek health services at MCH center.

Exclusion Criteria:

* single women not previously married
* and women who were married since more than one year

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Data will be collected through a semi-structured interviewer administered questionnaire Interviewer administered questionnaire
  1. Personal and demographic characters of women and their husbands; age, religion, current residence and residence in childhood (urban and rural), education, employment.
  2. Family characteristics: family type nuclear or extended, if the couples are blood relatives or not, media exposure, and assessment of family socioeconomic status using family income in L.E per month, response to the absence of economic difficulty in making it to the end of the month (much difficulty, difficulty, certain difficulty, much ease, ease, or certain ease)(10), and the Egypt socioeconomic scale by El-Gilany A (11).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
level of acceptability of intimate partner violence among ever married women | 2 years
  Acceptability to IVP will be measured using the A-IPVAW scale is a 20-item measure assessing attitudes of acceptability or tolerance of IPVAW (e.g., "It is acceptable for a man to shout at his partner if she is continuously arguing and nagging him, to hit his partner if she is constantly nagging/arguing, to push his partner into having sex because he spent money on her , to threaten to leave his partner in order to achieve something he wants, not to allow his partner to work or study, to prevent his partner from seeing family and friends, to control his partner's mobile phone"). The response format of these items is a 3-point Likert-type scale (i.e., 0 = "Not acceptable," 1 = "Somewhat acceptable," 2 = "Acceptable").

SECONDARY OUTCOMES:
level of victim blaming attitude in case of intimate partner violence | 2 years
  Victim-blaming attitudes in Cases of Intimate Partner Violence will be assessed using a short version of (VB-IPVAW). It composes of 12 items e.g.( men are violent towards their partners because they make them jealous, men are violent towards their partners because women provoke them, men are violent towards their partners because women need to be controlled, men are violent towards their partners because women are not patient enough with them, men would change their violent behavior towards their partners if they were more obedient, women could avoid violence from their malepartners if they knew when to stop talking). Respondents will be asked to indicate their level of agreement with the item statements on a 4-point Likert-type scale (1 = strongly disagree, 2= somewhat disagree, 3= somewhat agree, 4 = strongly agree).